CLINICAL TRIAL: NCT00436982
Title: Evaluation of Triathlon - a New Total Knee Prosthesis System. Prospective, Comparative, Randomised, Roentgen Stereophotogrammetric Analysis (RSA) Series
Brief Title: Evaluation of Triathlon - a New Total Knee Prosthesis System - Triathlon vs. Duracon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-S-015 Triathlon RSA_1; K-S-015_1 (Other: StrykerEuropean)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2015-12-08 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented Triathlon total knee system (Active Comparator): The Triathlon total knee system is the successor of the Duracon total knee system and was observed in a prospective randomised, parallel, double-blind study.
  Interventions: Device: Cemented Triathlon total knee system
- Cemented Duracon total knee system (Active Comparator): The Duracon total knee system is the predecessor of the Triathlon total knee system and was observed in a prospective randomised, parallel, double-blind study.
  Interventions: Device: Duracon total knee system

INTERVENTIONS:
Device: Cemented Triathlon total knee system — Orthopaedic implant
  Arms: Cemented Triathlon total knee system
Device: Duracon total knee system — Orthopaedic implant
  Arms: Cemented Duracon total knee system

SUMMARY:
The objective is to investigate the Clinical, Radiographic, Roentgen Stereophotogrammetric behaviour and patient outcome when using the Triathlon total knee prosthesis in a prospective randomized clinical trial.

DETAILED DESCRIPTION:
The evaluation is carried out by a prospective randomised RSA-study with Triathlon cemented knee prosthesis versus Duracon cemented knee prosthesis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suffering exclusively from osteo arthritis (OA), Stage II-V [Ahlbäck, 1968] will be operated.
2. Patients requiring knee prosthesis, suitable for the use of Duracon and Triathlon knee system
3. Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographical evaluations and the prescribed rehabilitation.
4. Patients who signed the Ethics Committee approved Informed Consent Form prior to surgery.

Exclusion Criteria:

1. Previous major knee surgery
2. Other significant disabling problems from the muscular-skeletal system than in the knees
3. Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI above 35).
4. Patients with active or suspected infection.
5. Patients with malignancy - active malignancy.
6. Patients with severe osteoporosis, Paget's disease, renal osteodystrophy.
7. Patients immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
8. The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
9. Female patients planning a pregnancy during the course of the study.
10. Patients with systemic or metabolic disorders leading to progressive bone deterioration.
11. Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
12. Patients with other severe concurrent joint involvements, which can affect their outcome.
13. Patients with other concurrent illnesses, which are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus or renal disease requiring dialysis.
14. Patients under the protection of law (e.g. guardianship).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-02; Primary Completion 2008-11 (Actual); Study Completion 2017-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sören Toksvig-Larsen, ass. prof, Principal Investigator — Department of ortopaedics, Hässleholm Hospital
Locations (1):
- Hässleholm Hospital, Hässleholm, Sweden

REFERENCES:
- [Result] Molt M, Ljung P, Toksvig-Larsen S. Does a new knee design perform as well as the design it replaces? Bone Joint Res. 2012 Dec 1;1(12):315-23. doi: 10.1302/2046-3758.112.2000064. Print 2012 Dec. PMID 23610663
- [Derived] Molt M, Toksvig-Larsen S. Similar early migration when comparing CR and PS in Triathlon TKA: A prospective randomised RSA trial. Knee. 2014 Oct;21(5):949-54. doi: 10.1016/j.knee.2014.05.012. Epub 2014 Jun 7. PMID 24974301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from February to November 2006. In a single centre patients were prospectively randomised to receive either a cemented Triathlon total knee system or a Duracon total knee system. Randomisation with envelopes, 30 patients in each group. Only one knee per participant was enrolled for the study.
Groups:
- Cemented Triathlon Total Knee System: 30 patients were randomized into the Triathlon total knee system arm. TheTriathlon total knee system is the successor of the Duracon total knee system and was observed in a prospective randomised, parallel, double-blind study.
  Cemented Triathlon total knee system: Orthopaedic implant
- Duracon Total Knee System: 30 patients were randomized into the Duracon total knee system arm. The Duracon total knee system is the predecessor of the Triathlon total knee system and was observed in a prospective randomised, parallel, double-blind study.
  Duracon total knee system: Orthopaedic implant
Period: Overall Study
Arm/Group | Cemented Triathlon Total Knee System | Duracon Total Knee System
Started | 30 | 30
Completed (Completed/Not completed counts based on participants status at the 2 year primary outcome interval) | 26 | 26
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Did not receive allocated intervention | 0 | 1
Not completed — no RSA data | 1 | 2

BASELINE CHARACTERISTICS:
Population: With an alpha of 0.05 and a beta of 0.20 the required sample size in each group is 25 patients to detect a difference of 0.3 mm. Patients with inadequate marking will be excluded from the study. Taking the latter into account and to compensate for possible lost to follow up, 30 patients will be recruited per study group.
Groups:
- Triathlon: 30 patients randomized into the Triathlon arm
- Duracon: 30 patients randomized into the Duracon arm
- Total: Total of all reporting groups
Arm/Group | Triathlon | Duracon | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Full Range); unit: years] | 69 [47 to 86] | 66 [47 to 84] | 68 [47 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 18 | 40
  Male | 8 | 12 | 20
Region of Enrollment [Number; unit: participants]
  Sweden | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Roentgen Stereophotogrammetric Analysis (RSA)
Description: To compare the maximum total point motion (MTPM) of the Triathlon and Duracon tibial components at two years assessed by means of RSA.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Triathlon | Duracon
Number analyzed (Participants) | 26 | 26
mm | 0.65 (0.66) | 0.81 (0.48)

2. Secondary Outcome: Roentgen Stereophotogrammetric Analysis (RSA)
Description: To compare the maximum total point motion (MTPM) of the Triathlon and Duracon tibial components by means of RSA.
Time Frame: 3 months, 1, 5, 7 and 10 years
Population: Participants with data available at each time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cemented Triathlon Total Knee System | Duracon Total Knee System
Number analyzed (Participants) | 30 | 30
mm
  MTPM 3 months: number analyzed (Participants) | 29 | 27
  MTPM 3 months | 0.45 (0.28) | 0.44 (0.27)
  MTPM 1 year: number analyzed (Participants) | 29 | 26
  MTPM 1 year | 0.6 (0.5) | 0.64 (0.36)
  MTPM 5 years: number analyzed (Participants) | 22 | 23
  MTPM 5 years | 0.65 (0.38) | 1.1 (1.19)
  MTPM 7 years: number analyzed (Participants) | 17 | 15
  MTPM 7 years | 0.67 (0.46) | 0.65 (0.3)
  MTPM 10 years: number analyzed (Participants) | 14 | 15
  MTPM 10 years | 0.75 (0.54) | 0.6 (0.28)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With KSS (Knee Society Score)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, ROM and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: [Time Frame: pre-operative, 3 months, 1, 2, 5, 7 and 10 years]
Population: Participants with data available at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Triathlon | Duracon
Number analyzed (Participants) | 30 | 30
units on a scale
  KSS Pain/Motion pre-operative | 17.3 (10.50) | 18.3 (11.24)
  KSS Pain/Motion 3 months: number analyzed (Participants) | 28 | 29
  KSS Pain/Motion 3 months | 86.09 (9.61) | 86.55 (14.57)
  KSS Pain/Motion 1 year: number analyzed (Participants) | 29 | 28
  KSS Pain/Motion 1 year | 93.51 (6.94) | 95.43 (9.71)
  KSS Pain/Motion 2 years: number analyzed (Participants) | 27 | 28
  KSS Pain/Motion 2 years | 94.96 (7.58) | 94.79 (7.55)
  KSS Pain/Motion 5 years: number analyzed (Participants) | 21 | 21
  KSS Pain/Motion 5 years | 93.14 (9.12) | 94.24 (9.71)
  KSS Pain/Motion 7 years: number analyzed (Participants) | 18 | 16
  KSS Pain/Motion 7 years | 90.06 (11.29) | 95.13 (11.21)
  KSS Pain/Motion 10 years: number analyzed (Participants) | 15 | 16
  KSS Pain/Motion 10 years | 93.6 (10.45) | 96.79 (6.83)
  KSS Function pre-operative | 51.17 (12.30) | 53.67 (6.81)
  KSS Function 3 months: number analyzed (Participants) | 28 | 29
  KSS Function 3 months | 70 (10.89) | 72.76 (14.91)
  KSS Function 1 year: number analyzed (Participants) | 29 | 26
  KSS Function 1 year | 80 (18.17) | 84.42 (15)
  KSS Function 2 years: number analyzed (Participants) | 27 | 28
  KSS Function 2 years | 86.67 (14.9) | 88.57 (15.51)
  KSS Function 5 years: number analyzed (Participants) | 22 | 21
  KSS Function 5 years | 81.82 (20.68) | 81.67 (18.66)
  KSS Function 7 years: number analyzed (Participants) | 18 | 16
  KSS Function 7 years | 76.11 (27.73) | 92.5 (15.71)
  KSS Function 10 years: number analyzed (Participants) | 15 | 16
  KSS Function 10 years | 78.33 (21.10) | 84.38 (16.82)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With KOOS Patient Questionnaire
Description: KOOS consists of 5 subscales; Pain, other Symptoms, Activities of Daily Living (ADL), Sport and Recreation Function (Sport/Rec) and knee-related Quality of Life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
  [taken from User Guide] http://www.koos.nu/
Time Frame: pre-operative, 3 months, 1, 2, 5, 7 and 10 years
Population: Participants with data available at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cemented Triathlon Total Knee System | Duracon Total Knee System
Number analyzed (Participants) | 30 | 30
units on a scale
  QOL pre-operative | 23.75 (14.44) | 24.38 (14.62)
  QOL 3 months: number analyzed (Participants) | 28 | 29
  QOL 3 months | 51.79 (20.61) | 54.09 (23.87)
  QOL 1 year: number analyzed (Participants) | 28 | 27
  QOL 1 year | 58.48 (22.13) | 65.51 (21.04)
  QOL 2 years: number analyzed (Participants) | 27 | 28
  QOL 2 years | 62.73 (25.56) | 71.35 (25.42)
  QOL 5 years: number analyzed (Participants) | 22 | 21
  QOL 5 years | 69.87 (30.04) | 80.06 (18.71)
  QOL 7 years: number analyzed (Participants) | 18 | 16
  QOL 7 years | 68.75 (28.36) | 86.33 (12.95)
  QOL 10 years: number analyzed (Participants) | 15 | 17
  QOL 10 years | 65.83 (25.1) | 73.53 (27.56)
  Symptoms preoperative | 51.25 (18.67) | 53.65 (16.36)
  Symptoms 3 months: number analyzed (Participants) | 28 | 29
  Symptoms 3 months | 66.84 (18.62) | 65.87 (17.50)
  Symptoms 1 year: number analyzed (Participants) | 28 | 27
  Symptoms 1 year | 75.51 (17.08) | 77.51 (15.84)
  Symptoms 2 years: number analyzed (Participants) | 27 | 28
  Symptoms 2 years | 78.17 (16.29) | 81.87 (16.57)
  Symptoms 5 years: number analyzed (Participants) | 22 | 21
  Symptoms 5 years | 81.81 (20.41) | 83.16 (19.40)
  Symptoms 7 years: number analyzed (Participants) | 17 | 16
  Symptoms 7 years | 82.14 (15.87) | 92.63 (14.13)
  Symptoms 10 years: number analyzed (Participants) | 15 | 17
  Symptoms 10 years | 81.62 (19.15) | 88.45 (13.15)
  Pain preoperative | 42.11 (16.88) | 43.61 (14.07)
  Pain 3 months: number analyzed (Participants) | 28 | 29
  Pain 3 months | 70.57 (20.23) | 70.21 (21.52)
  Pain 1 year: number analyzed (Participants) | 28 | 27
  Pain 1 year | 73.64 (19.39) | 82.77 (19.59)
  Pain 2 years: number analyzed (Participants) | 27 | 28
  Pain 2 years | 79.94 (19.89) | 84.82 (20.83)
  Pain 5 years: number analyzed (Participants) | 22 | 21
  Pain 5 years | 81.31 (21.23) | 85.45 (19.44)
  Pain 7 years: number analyzed (Participants) | 18 | 16
  Pain 7 years | 80.56 (19.29) | 91.15 (14.74)
  Pain 10 years: number analyzed (Participants) | 15 | 17
  Pain 10 years | 80.74 (19.20) | 84.31 (20.99)
  ADL preoperative | 47.27 (14.58) | 50.14 (15.58)
  ADL 3 months: number analyzed (Participants) | 28 | 29
  ADL 3 months | 73.22 (18.23) | 73.35 (23.09)
  ADL 1 year: number analyzed (Participants) | 28 | 27
  ADL 1 year | 74.28 (20.23) | 84.42 (15.45)
  ADL 2 years: number analyzed (Participants) | 27 | 28
  ADL 2 years | 76.74 (21.78) | 84.90 (20.22)
  ADL 5 years: number analyzed (Participants) | 22 | 21
  ADL 5 years | 78.07 (23.60) | 83.05 (19.39)
  ADL 7 years: number analyzed (Participants) | 18 | 16
  ADL 7 years | 75.25 (22.90) | 89.34 (13.18)
  ADL 10 years: number analyzed (Participants) | 14 | 17
  ADL 10 years | 73.21 (24.42) | 80.02 (24.98)
  Sport/Rec preOP | 6.5 (8.22) | 10 (14.20)
  Sport/Rec 3 months: number analyzed (Participants) | 27 | 28
  Sport/Rec 3 months | 20.19 (18.58) | 29.55 (21.50)
  Sport/Rec 1 year: number analyzed (Participants) | 27 | 26
  Sport/Rec 1 year | 30.46 (23.80) | 38.65 (28.52)
  Sport/Rec 2 years: number analyzed (Participants) | 26 | 27
  Sport/Rec 2 years | 28.65 (21.66) | 46.17 (32.47)
  Sport/Rec 5 years: number analyzed (Participants) | 22 | 21
  Sport/Rec 5 years | 36.14 (26.50) | 38.33 (30.51)
  Sport/Rec 7 years: number analyzed (Participants) | 18 | 16
  Sport/Rec 7 years | 22.5 (25.34) | 44.06 (33.08)
  Sport/Rec 10 years: number analyzed (Participants) | 15 | 17
  Sport/Rec 10 years | 25.33 (19.68) | 50.15 (30.29)

5. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With EQ-5D Patient Questionnaire
Description: The EQ-5D is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; the EQ visual analogue scale (EQ VAS) and EQ-5D descriptive system. The EQ VAS collects health state values using a 20 cm visual analogue scale with the endpoints labeled best imaginable health state at the top and worst imaginable health state at the bottom, having numeric values of 100 to 0 respectively. The EQ-5D Time Trade-off (TTO) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/comfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems, where an overall score of 1 represents full health.
  NOTE: While the protocol includes pre-operative, 3 months, and 1 year, this data was not collected.
Time Frame: pre-operative, 3 months, 1, 2, 5, 7 and 10 years
Population: Participants with data available at each time point. Overall number of participants and units analyzed is based upon the 2 year population
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Triathlon Total Knee System: 30 patients were randomized into the Duracon total knee system arm. The Duracon total knee system is the predecessor of the Triathlon total knee system and was observed in a prospective randomised, parallel, double-blind study.
  Triathlon total knee system: Orthopaedic implant
Arm/Group | Duracon Total Knee System | Triathlon Total Knee System
Number analyzed (Participants) | 28 | 26
units on a scale
  EQ-5D 2 years | 0.79 (0.24) | 0.80 (0.22)
  EQ-5D 5 years: number analyzed (Participants) | 21 | 22
  EQ-5D 5 years | 0.76 (0.30) | 0.78 (0.26)
  EQ-5D 7 years: number analyzed (Participants) | 16 | 18
  EQ-5D 7 years | 0.86 (0.24) | 0.73 (0.29)
  EQ-5D 10 years: number analyzed (Participants) | 17 | 15
  EQ-5D 10 years | 0.78 (0.24) | 0.75 (0.26)

6. Secondary Outcome: Mean Operative Time
Description: Skin to skin operative time
Time Frame: intra-operative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Triathlon | Duracon
Number analyzed (Participants) | 30 | 30
minutes | 66.47 (9.62) | 63.7 (12.21)

7. Secondary Outcome: Duration Hospital Stay
Time Frame: preoperative to discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Triathlon | Duracon
Number analyzed (Participants) | 30 | 30
days | 4.9 (2.58) | 4.76 (0.91)

8. Secondary Outcome: Blood Loss
Description: Blood loss during surgery
Time Frame: intra-operative
Population: The protocol indicates blood loss as a secondary measure but this value was not collected. Therefore no data can be posted.
Arm/Group | Triathlon | Duracon
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: During entire 10 years follow-up of all patients
Description: All serious adverse events and operative site events occuring in this study were reported.
Arm/Group | Triathlon | Duracon
Serious Adverse Events (participants affected / at risk) | 4/30 | 3/30
Other Adverse Events (participants affected / at risk) | 4/30 | 5/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon (N=30) | Duracon (N=30)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
Fracture proximal tibia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hip fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Supercondylar humerus fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triathlon (N=30) | Duracon (N=30)
Deep Vein Thrombosis (Vascular disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less